CLINICAL TRIAL: NCT06986005
Title: Investigation of the Effect of Neoadjuvant Chemotherapy on Physical Functions in Women With Breast Cancer
Brief Title: The Effect of Neoadjuvant Chemotherapy on Physical Functions
Status: Recruiting | Type: Observational
Sponsor: ATİYE KAŞ ÖZDEMİR (Other)
Responsible Party: Sponsor-Investigator, ATİYE KAŞ ÖZDEMİR, Lecturer PhD., Pamukkale University
Organization: Pamukkale University (Other)
Other Study IDs: E-60116787-020-642610
Record Dates: First submitted 2025-05-04; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer; Neoadjuvant Chemotherapy; Neoadjuvant Therapy
Keywords: physical functions; breast cancer; neoadjuvant chemotherapy; physiotherapy; fatigue; physical activity
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Breast cancer patients receiving neoadjuvant chemotherapy: Breast cancer patients who receiving neoadjuvant chemotherapy
  Interventions: Other: No intervention will be performed as part of this study. However, regardless of the study, all participants will receive neoadjuvant chemotherapy.

INTERVENTIONS:
Other: No intervention will be performed as part of this study. However, regardless of the study, all participants will receive neoadjuvant chemotherapy. — All participants will receive neoadjuvant chemotherapy appropriate to the characteristics of their breast cancer as part of their standard care.

SUMMARY:
The aim of this observational study was to investigate the effect of neoadjuvant chemotherapy on physical functioning in individuals with breast cancer. The main question that the study aims to answer is how the physical functions of individuals are after neoadjuvant chemotherapy. Demographic information of the participants will be recorded and their physical status will be evaluated by determining body weight and composition, 30-second sit-and-stand test, 9-step stair ascent and descent test, one-leg stand test, upper extremity muscle strength test, lower extremity muscle strength test, tissue dielectric constant measurement, Lower Extremity Functional Scale, Global Physical Activity Questionnaire and Multidimensional Fatigue Rating Scale. In these patients who are planned to receive neoadjuvant chemotherapy for breast cancer, measurements will be made before chemotherapy (T1) and after chemotherapy (T2).

DETAILED DESCRIPTION:
As a result of the power analysis made from the reference study; when the effect size d=0.8, it was calculated that 80% power could be obtained at 95% confidence level when at least 42 people were included in the study. Considering that a lower effect size can also be obtained, it is planned to complete the study with at least 46 participants by taking 10% more participants.

The data will be analysed with SPSS 25.0 package programme. Continuous variables will be given as mean ± standard deviation and categorical variables as number and percentage. When parametric test assumptions are met, the Significance Test of the Difference Between Two Means will be used to compare independent group differences; when parametric test assumptions are not met, the Mann-Whitney U test will be used to compare independent group differences. In dependent group comparisons, repeated measures analysis of variance will be used when parametric test assumptions are met; Friedman test will be used when parametric test assumptions are not met. In addition, the relationships between continuous variables will be examined by Spearman or Pearson correlation analyses and the differences between categorical variables will be examined by Chi-square analysis.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are planned to receive neoadjuvant chemotherapy for breast cancer
* Acceptance to participate in the study

Exclusion Criteria:

* Previous history of breast cancer
* History of any other cancer
* Refusal to participate in the study
* Refusal to continue working

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Individuals who are followed up by Pamukkale University Breast Polyclinic
Sampling Method: Non-Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Upper limb muscle strength | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  Since hand grip strength is correlated with upper extremity muscle strength as well as general body muscle strength and pulmonary muscle strength, upper extremity muscle strength will be evaluated by hand dynamometer.
Lower limb muscle strength | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  Lower extremity muscle strength will be measured with Hand Held Dynamometer.
9 stair ascent and descent test | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  A 9-step stair ascent and descent test will be used to assess the patient's stair ascent and descent activity, dynamic balance and lower extremity strength.
Balance assessment | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  Balance will be assessed in two stages: static and dynamic balance. Standing on one leg test will be used as static balance assessment and 30 seconds sit-and-stay test will be used for dynamic balance assessment.
Lower Extremity Function | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  The Lower Extremity Functional Scale developed by Binkley et al. (1999) to evaluate lower extremity function, activity limitations of individuals, lower extremity functions and abilities in patients with musculoskeletal disorders will be used.

SECONDARY OUTCOMES:
Physical activity level | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  The Global Physical Activity Questionnaire, which is a self-report form consisting of 16 questions prepared by the World Health Organisation (WHO), will be used.
Fatigue | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  The Multidimensional Fatigue Rating Scale will be used to measure the fatigue levels of the participants.
Determination of body weight and composition | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  The weight of the participants will be measured directly with a Tanita device that works with the segmental multi-frequency bioelectrical impedance analysis method. The Tanita Bady Fat Monitor works with the Bioelectrical Impedance Analysis technique. This method analyses the composition of the body. An imperceptible, very weak and body-safe electric current circulates in the fluid inside the muscles. When the current encounters the fat layer, it encounters resistance, the layers showing resistance are evaluated by the device, compared with weight and height and displayed on the digital screen as fat ratio.
Tissue dielectric constant measurement | It is planned to repeat the measurements 2 times: baseline and after the procedure ofneoadjuvant chemotherapy.
  Subdermal fluid measurements by tissue dielectric constant are one of the best methods to diagnose and localise early lymphoedema and also to identify a number of non-lymphoedema patients potentially at risk for later lymphoedema formation. Tissue dielectric constant will be determined by measuring the sub-tissue fluid density of the individuals at defined reference points using a Moisture Meter-D compact (MMDc, Delfin Technologies, Finland).

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No